CLINICAL TRIAL: NCT06809101
Title: Home Monitoring of Complete Blood Count Performed by Patients - a Pilot Study on the Implementation Process in South Baltic Countries.
Acronym: AMBeR eBlood
Status: Recruiting | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: University Clinical Centre, Gdansk (Other); University Medicine Greifswald (Other); University Medical Center Rostock (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: p-2024-17504; STHB.01.01-IP.01-0005/23 (Other Grant/Funding Number: Interreg South Baltic 2021-2027 programme)
Record Dates: First submitted 2025-01-18; First posted 2025-02-05 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Cancer-related Problem/Condition; Chemotherapy; Chemotherapy-induced Neutropenia; Chemotherapy Induced Anaemia; Chemotherapy Induced Thrombocytopenia
Keywords: home blood monitoring; complete blood count; cancer; chemotherapy; implementation; research; e-health; oncology; home-based; feasibility
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Oncology patients undergoing home blood monitoring. n=33 per site.
- Control group: Oncology patients undergoing standard blood testing in the general laboratory at the Outpatient Clinic.
  n=20 per site.

SUMMARY:
Introduction:

The number of diagnosed cancers is systematically increasing every year. Cancer patients need to undergo regular blood tests to monitor safety and eligibility for treatment. In case of poor blood results, the chemotherapy session must be omitted. For patients living far from the center, this means unnecessary travel with involvement of helpers, additional costs, increased potential of hospital acquired infections, and frustration associated with missed opportunity for treatment.

Aims:

The primary aim of this study is to gain knowledge about successful implementation of remote, home monitoring of complete blood count to cancer patients during and after systemic treatment for cancer. The secondary aim of the AMBeR collective study protocol is to pilot new technology, gain more context around future investigations and verify costs and changes in patient treatment pathways.

Methodology:

The investigators will test implementation of home blood monitoring in three South Baltic Countries (DK, PL, GER). Each site will participate in the implementation study with study group á n=33 (total n=165) and control group n=20 (total n=100). The duration of the study is planned for 4 cycles of chemotherapy for each patient and a 3-month follow up period. The ﬁrst cycle of learning and training at the Outpatient Daily Clinic, then the remaining 3 cycles of blood monitoring at home. The average cycle length is 21-30 days, number of measurements will be determined individually depending on the diagnosis. At a baseline, after 4 cycles of chemotherapy (12-16 weeks) and after a 3-month follow-up period, parallel studies will be carried out in both the study and control groups, using mixed methods the investigators will assess outcomes of reach, effectiveness, adoption, implementation and maintenance (RE-AIM).

Expected beneﬁts:

Implementation of the AMBeR study should reduce the amount of unnecessary and nontherapeutic hospital visits and improve manageability and independence of the patients. The investigators believe that the decrease in the number of hospital visits will diminish the risk of infection for vulnerable individuals, as well as save costs for patients and hospitals. These factors will also translate into better logistics of chemotherapy units, decreased carbon-dioxide trail, and improved quality of life and patient empowerment.

DETAILED DESCRIPTION:
Introduction:

The incidence of cancer is expected to increase by 30% over the next 20 years, mainly due to the increase in the elderly population. This will lead to a dramatic increase in the number of cancer patients in the future. Cancer patients need to undergo regular blood tests to monitor safety and eligibility for treatment. In case of poor blood results, the chemotherapy session must be omitted or modified. For patients living far from the center, this means unnecessary travel with involvement of helpers, additional costs, increased potential of hospital acquired infections, and frustration associated with missed opportunity for treatment. Digitizing cancer care can increase patients' active involvement in their own treatment, improve quality of life and reduce inequalities in access to health care. Therefore, there is a strong need to develop and implement new ways of making cancer diagnostics and treatments available to patients in their own homes.

Objective The primary aim of this study is to gain knowledge about successful implementation of remote, home monitoring of complete blood count to cancer patients during systemic treatment for cancer. The secondary aim of the AMBeR collective study protocol is to pilot new technology, gain more context around future investigations and verify costs and changes in patient treatment pathways.

Methods

Trial design This study is a multinational multisite implementation research study to pilot test implementation of home blood monitoring in 3 South Baltic countries (PL, DK, GER).

Study setting and organization The current study is part of the Interreg South Baltic Program-funded project "AMBeR" (Advanced Modelling of Baltic cancer e-caRe). A total of seven partners from five countries are involved and are working on five different WP's. The following 5 of the 7 project partners are involved in the study (WP3): 1) Zealand University Hospital Næstved, Denmark (ZUH); 2) University Medical Center Rostock, Germany (UMC Rostock); 3) University Medical Center Greifswald, Germany (UMC Greifswald); 4) University Clinical Center Gdańsk, Poland (UCC Gdańsk); 5) Pomeranian Medical University Szczecin, Poland (PMU).

Intervention The aim of this study is to evaluate the feasibility and validity of home monitoring of blood parameters during systemic treatment of cancer patients using the HemoScreen device in the patient's home. Participants will be oncology patients undergoing outpatient chemotherapy in Oncology and Hematology Departments in 5 different centers in the South Baltic region.

The investigators plan to enroll 33 patients from each center in the study group and 20 patients in the control group. Patients in the control group will undergo standard chemotherapy treatment and blood monitoring in general laboratory at the Outpatient Daily Clinic.

Patients from the study group will be instructed in the use of the HemoScreen device by trained staff and will complete self-tests throughout their first cycle of chemotherapy at the Outpatient Daily Clinic (average cycle duration 21-30 days, number of measurements determined individually depending on the diagnosis). Patients will then be given HemoScreen to use at home and will be tested immediately or up to 48 hours before their scheduled outpatient visit for chemotherapy. The results obtained will be sent to the coordinator via the IT system at least 24 hours before the planned administration of chemotherapy to determine contraindications to treatment.

If the results do not qualify for chemotherapy, depending on the center, a decision will be made to arrive to the Outpatient Daily Clinic to verify the test or to postpone the visit and issue recommendations. Each time a patient arrives at the Outpatient Day Clinic for chemotherapy, a standard venous blood test will be performed in the general laboratory. Any decision on the final administration of chemotherapy will be based on the blood count obtained from the general laboratory, not from the HemoScreen device. All trial procedures are done in addition to standard care.

The duration of the study was planned for 4 cycles of chemotherapy for each patient and a 3-month follow-up period. The first cycle of learning and training at the Outpatient Daily Clinic, then the remaining 3 cycles of blood monitoring at home. At a baseline, after 4 cycles of chemotherapy (12-16 weeks) and after a 3-month follow-up period, parallel studies will be carried out in both the study and control groups, using questionnaires (PROM's) assessing a health status and quality of life to evaluate the impact of an intervention.

Implementation

* describing the existing care process and identifying stakeholders.
* describing new care process, stakeholders and pathways in the new practice.
* Workshop 1:" setting the scene" context mapping, barriers and facilitators, solution design, action plan. Participation from all relevant stakeholders identified through context mapping of the care process. A patient representative will be involved and engaged in workshop if possible, and thereby contribute with the patient perspective on barriers and facilitators.
* Education and preparing health care professionals (HCP's) to use of the digital technology and integrating it into the "toolbox" and new professional identity.
* Workshop 2 "facilitating/supporting the ongoing process" mid-pilot, dealing with challenges, adjusting design, planning, and supporting further implementation.
* Workshop 3 "selecting the fruits of best practice" post-pilot, including examining learnings from the pilot trials and evaluating finalized, ongoing and planned implementation.
* A logbook describing the process, actions, and rationale for all steps of the implementation will be used for documentation throughout the intervention phase.

Following workshop 1, pre-study identification of expected barriers and facilitators for patients to engage in remote blood monitoring at home will be carried out in 4 steps:

* Summary from literature review and past experiences.
* Matching the most important barriers with strategies using the ERIC matching tool.
* Ranking strategies by effectiveness and importance in each center's clinical setting.
* Building on strategies to develop action plans to implement interventions in each site.

Assessing RQ1: Patient's and HCP's perspectives on determinants

In the final phase of the pilot study, the investigators will examine the perspectives of patients and HCPs on important determinants of engagement in remote home blood monitoring using the Group Concept Mapping technique. The process will follow 5 pre-described steps and all activity will be online utilizing the software Groupwisdom:

1. Brainstorming
2. Sorting and labelling
3. Rating
4. Generating a cluster rating map
5. Validation of the cluster rating map

Quantitative outcomes The investigators will use the RE-AIM framework (REF) for a systematic quantification of outcomes. A range of different outcomes, measurement methods and data sources will be used.

Data collection and management A REDCap database will be created for all study outcomes and relevant data to be collected and safely stored.

Participant and Non-participant questionnaires To obtain information about eligible patients who refuse participation in remote home blood monitoring, the investigators will invite patients to complete a short survey containing information about their characteristics, reasons for refusal, and barriers to participation. Patients who accept participation will receive a larger questionnaire reporting further on Patient Reported Outcome Measures (PROMs) and Patient Reported Experience Measures (PREMs). PROMs and PREMs will be collected using validated questionnaires. Additionally, the investigators want to examine the implementation process. To this end, a survey will be conducted at the end of the study to examine participants' and medical professionals' experiences of implementation.

Effectiveness evaluation At the baseline, after 16 weeks of treatment and 3 months of follow-up, a survey will be conducted regarding patients' perceptions of their care experience, including quality of life (PROM's - EORTC QLQ C30; EQ-5D 5L) and acceptability (Theoretical framework of Acceptability). Adherence to home blood testing and adverse events will be recorded throughout the study. At the same time, the investigators will analyze the number of unnecessary and non-therapeutic hospital visits that could potentially be avoided. Finally, health economic data will be collected to assess the economic value of the project and conduct cost-benefit analysis.

Harms and drop-outs Remote blood monitoring may be associated with adverse events and the ongoing and systematic registration of harm, drop-out and reasons for drop-out. This information will be recorded in the database on a day-to-day basis.

Economic/resource evaluation Based on the collected process data, the investigators will conduct an economic analysis assessing the time, resources and costs used for remote home monitoring. Additionally, the investigators would like to evaluate the price of the device with disposable materials, maintenance costs, time and amount of money necessary for training. Thanks to the above calculations, the investigators will try to estimate the cost-effectiveness of the change and the effective use of resources to perform blood test at home.

Sample size in pilot trials First, sample size of the pilot trial was estimated based on considerations to ensure sufficient accumulation of experience at each site to draw upon in the development of eMOC, supported by the literature on sample size recommendations for pilot and feasibility trials.

Second, the investigators defined success in the study if patients were able to use the HemoScreen equipment properly at home by following the instructions they received. Failure was defined as when the patients must call the helpline or notice that they are not using the equipment correctly at home. The investigators assumed the expected probability of success at po = 0.90. The investigators decided that if the probability of success is p=0.70 (or less), then the HemoScreen may not be useful in a given context. The null hypothesis of the study is Ho: p = p0, and the investigators wanted to test the alternative hypothesis Ha: p <p0 (one-tailed test) with a probability of 5% or less and a power of 80%. The estimated necessary sample size is N = 33 patients.

By consortium decision, each pilot study included 33 participants at each site, resulting in a total pooled sample of 165 participating patients. The consortium decided to enroll 20 control patients from each site, resulting in a total sample of 100 participants. Therefore, a total of 265 patients were planned to participate in the entire study.

Statistical methods Mainly descriptive statistics will be used to analyze quantitative outcomes, although effectiveness will be assessed with a pre-post change score.

Ethics approval and consent to participate An application for ethics approval will be submitted in each participating country, with local adaptations of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* legally competent patients
* aged 18 or older
* diagnosed with cancer (ICD-10: C00* - C97*)
* enrolled at the Department of Oncology/Hematology for outpatients
* participants who are willing and able to give informed consent for participation in the study
* participants should receive chemotherapy in Daily Chemotherapy Unit and be within 4 weeks of chemotherapy initiation, and the expected duration of chemotherapy should be at least 12 weeks from inclusion

Exclusion Criteria:

* inability to give informed consent due to mental capacity or language barrier
* patient unable or unlikely to be able to perform fine manipulation required to use lancet or cartridge to obtain capillary blood sample and result
* known bleeding disorder
* bad circulation preventing the patient from getting enough blood drops to perform the test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are patients that suffer from cancer, require outpatient chemotherapy, and have sufficient manual skills and good eyesight to independently perform home blood monitoring, and sufficient cognitive skills to operate POCT and transfer data.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Patient's perspectives on determinants assessed by Group Concept Mapping | from 4 to 12 weeks of patient participation in the intervention
  Following completion or in the final phase of the pilot study, the investigators will examine the perspectives of patients on important determinants of engagement in remote home blood monitoring using the Group Concept Mapping technique. The process will follow 5 pre-described steps and all activity will be online utilizing the software Groupwisdom. The steps are as follows:
  1. Brainstorming
  2. Sorting and labelling
  3. Rating
  4. Generating a cluster rating map
  5. Validation of the cluster rating map
  The investigators will invite a representative sample of patients for study.

OTHER OUTCOMES:
Healthcare proffessionals' perspectives on determinants assessed by Group Concept Mapping | between 5 patient treatments completed and end of study (on average 1 year)
  Following completion or in the final phase of the pilot study, the investigators will examine the perspectives of HCPs on important determinants of engagement in remote home blood monitoring using the Group Concept Mapping technique. The process will follow 5 pre-described steps and all activity will be online utilizing the software Groupwisdom. The steps are as follows: 1) Brainstorming 2) Sorting and labelling 3) Rating 4) Generating a cluster rating map 5) Validation of the cluster rating map The investigators will invite all participating intervention delivering HCP´s to the study.
Number of referrals | Baseline
  Number of referred patients
Recruitment rates | Baseline
  Number of enrolled vs. declined
Sex of enrolled patients | Baseline
  a) male; b) female
Sex of decliners | Baseline
  a) male; b) female
Body height of enrolled patients | Baseline
  Measured in meters
Body height of decliners | Baseline
  Measured in meters
Body weight of enrolled patients | Baseline
  Measured in kilograms
Body weight of decliners | Baseline
  Measured in kilograms
Cancer disease of enrolled patients | Baseline
  Cancer type, cancer treatment, treatment intent
Cancer disease of decliners | Baseline
  Cancer type, cancer treatment, treatment intent
Educational level of enrolled patients according to International Standard Classification of Education | Baseline
  International Standard Classification of Education (ISCED) ISCED 0 = Early childhood education ISCED 1 = Primary Education ISCED 2 = Lower Secondary Education ISCED 3 = Upper Secondary Education ISCED 4 = Post-secondary non-Tertiary Education ISCED 5 = Short-cycle tertiary education ISCED 6 = Bachelors degree or equivalent tertiary education level ISCED 7 = Masters degree or equivalent tertiary education level ISCED 8 = Doctoral degree or equivalent tertiary education level
Educational level of decliners according to International Standard Classification of Education | Baseline
  International Standard Classification of Education (ISCED) ISCED 0 = Early childhood education ISCED 1 = Primary Education ISCED 2 = Lower Secondary Education ISCED 3 = Upper Secondary Education ISCED 4 = Post-secondary non-Tertiary Education ISCED 5 = Short-cycle tertiary education ISCED 6 = Bachelors degree or equivalent tertiary education level ISCED 7 = Masters degree or equivalent tertiary education level ISCED 8 = Doctoral degree or equivalent tertiary education level
Employment status of enrolled patients | Baseline
  a) Full time, b) part time, c) self-employed, d) unemployed seeking work, e) unemployed not seeking work, f) student, g) retired, h) unable to work, i) other
Employment status of decliners | Baseline
  a) Full time, b) part time, c) self-employed, d) unemployed seeking work, e) unemployed not seeking work, f) student, g) retired, h) unable to work, i) other
Distance to facility of enrolled patients | Baseline
  Measured in km
Distance to facility of decliners | Baseline
  Measured in km
Transport time to facility of enrolled patients | Baseline
  Measured in minutes
Transport time to facility of decliners | Baseline
  Measured in minutes
Health technology readiness assessed by Readiness and Enablement Index for Health Technology | Assessed pre-, post-intervention (16 weeks) and after 3 months of follow up
  The Readiness and Enablement Index for Health Technology (READHY) instrument consists of 13 dimensions with a total of 65 items. All 13 scales reflect the conceptual dimensions and are rated on a Likert-type scale from 1=strongly disagree to 4=strongly agree
European Organization of Research and Treatment in Cancer, core module (C30) | Assessed pre-, post-intervention (16 weeks) and after 3 months of follow up
  Health Related Quality of Life tool for use in clinical trials in oncology, consisting of 30 questions, from which one can obtain points from 0 to 100. The higher the score, the lower the patient's quality of life.
EuroQol-5 Dimensions-5 Levels | Assessed pre-, post-intervention (16 weeks) and after 3 months of follow up
  EuroQol-5 Dimensions-5 Levels (EQ-5D 5L) is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire. For the EQ-5D-5L questionnaire, 3125 health states were defined: from "11111" (no problems at all) to "55555" ("extreme problems" in all five domains)
Attendance rate | Assessed post-intervention (16 weeks)
  Number of home blood tests performed versus number of tests ordered
Adverse events during home blood testing | Assessed post-intervention (16 weeks)
  Registration of all adverse events throughout the intervention
Acceptability for patients assessed using the Theoretical Framework of Acceptability Questionnaire | Assessed post-intervention (16 weeks)
  Theoretical Framework of Acceptability (TFA) Questionnaire is used to assess operational problems and failure rates in terms of technology and language. It consists of 8 questions that can be answered on a scale of difficulty in using technology or understanding the language from 1 (min.) to 5 (max.).
Acceptability for healthcare professionals assessed using the Theoretical Framework of Acceptability Questionnaire | Assessed post-intervention (16 weeks)
  Theoretical Framework of Acceptability (TFA) Questionnaire is used to assess operational problems and failure rates in terms of technology and language. It consists of 8 questions that can be answered on a scale of difficulty in using technology or understanding the language from 1 (min.) to 5 (max.).
Administrative time consumption per patient | Assessed post-intervention (16 weeks)
  Measured in minutes and number of contact attempts
Medical time consumption per patient | Assessed post-intervention (16 weeks)
  Measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Bogusław Machaliński, MD, PhD, Prof, Principal Investigator — Department of Hematology and Transplantology, Pomeranian Medical University in Szczecin
Locations (5):
- Department of Oncology, Zealand University Hospital, Næstved, Region Sjælland, Denmark
- Germany (2):
  - Clinic and Polyclinic for Internal Medicine C, Hematology and Oncology, Palliative Care Unit, University Medical Center, Greifswald, Mecklenburg-Vorpommern
  - Department of Medicine, Clinic III, Hematology, Oncology, Palliative Medicine, University Medical Center, Rostock, Mecklenburg-Vorpommern
- Poland (2):
  - Department of Oncology and Radiotherapy, University Clinical Center of Gdańsk,, Gdansk, Pomeranian Voivodeship
  - Department of Hematology and Transplantology, Szczecin, West Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Homepage for the AMBeR project, of which the AMBeR Home Blood Monitoring is a work package and separately registered study. — https://amber.ku.lt/en/advanced-modeling-of-baltic-cancer-e-care-amber